CLINICAL TRIAL: NCT07352228
Title: Carvedilol vs. Propranolol for Preventing Rebleeding After Endoscopic Treatment of Cirrhotic Varices: A Single-Center Randomized Controlled Trial
Brief Title: Carvedilol vs. Propranolol for Preventing Rebleeding After Endoscopic Treatment of Cirrhotic Varices
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XJLL-KY-20252468
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Rebleeding of Portal Hypertension in Liver Cirrhosis; Propranolol; Carvedilol
MeSH Terms: interventions — Propranolol; Carvedilol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol group (Active Comparator): Oral carvedilol is administered within 24-72 hours after enrollment, with an initial dose of 6.25 mg once daily. After 3 days to 1 week, if systolic blood pressure ≥ 90 mmHg, heart rate ≥ 55 beats/min, and no significant adverse reactions, the dose is increased to 6.25 mg twice daily. If heart rate < 55 beats/min, systolic blood pressure < 90 mmHg, or significant adverse reactions occur, the dose is reduced to 6.25 mg once daily; intolerable cases discontinue medication and are recorded as adverse events. Maximum dose: 12.5 mg/day (25 mg/day may be considered for patients with persistent hypertension after physician evaluation, with close blood pressure monitoring). During the first 3 months of dose adjustment, heart rate and blood pressure are checked monthly; after dose stabilization, they are checked every 3 months. Medication adherence is monitored via telephone follow-up.
  Interventions: Drug: Carvedilol
- Propranolol Group (Placebo Comparator): Oral propranolol is administered within 24-72 hours after enrollment, with an initial dose of 10-20 mg twice daily. Heart rate is monitored 12-24 hours after medication initiation. Target heart rate: 50-60 beats/min or 75% of the baseline value. If the target heart rate is achieved without adverse reactions, the current dose is maintained. If not achieved without adverse reactions, the dose is gradually increased by 10-20 mg/day (divided into 2 doses; e.g., 20 mg/day can be increased to 30-40 mg/day, still twice daily). Maximum dose: 320 mg/day. If the maximum dose is reached without achieving the target heart rate, the maximum dose is maintained. If adverse reactions (e.g., bradycardia, hypotension) occur, the dose is immediately reduced to the maximum tolerated dose; intolerable cases discontinue medication and are recorded as adverse events. During the first 3 months of dose adjustment, heart rate is checked monthly; after dose stabilization, it is checked every 3 months.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Oral propranolol is administered within 24-72 hours after enrollment, with an initial dose of 10-20 mg twice daily. Heart rate is monitored 12-24 hours after medication initiation. Target heart rate: 50-60 beats/min or 75% of the baseline value. If the target heart rate is achieved without adverse reactions, the current dose is maintained. If not achieved without adverse reactions, the dose is gradually increased by 10-20 mg/day (divided into 2 doses; e.g., 20 mg/day can be increased to 30-40 mg/day, still twice daily). Maximum dose: 320 mg/day. If the maximum dose is reached without achieving the target heart rate, the maximum dose is maintained. If adverse reactions (e.g., bradycardia, hypotension) occur, the dose is immediately reduced to the maximum tolerated dose; intolerable cases discontinue medication and are recorded as adverse events. During the first 3 months of dose adjustment, heart rate is checked monthly; after dose stabilization, it is checked every 3 months.
  Other Names: inderol
  Arms: Propranolol Group
Drug: Carvedilol — Oral carvedilol is administered within 24-72 hours after enrollment, with an initial dose of 6.25 mg once daily. After 3 days to 1 week, if systolic blood pressure ≥ 90 mmHg, heart rate ≥ 55 beats/min, and no significant adverse reactions, the dose is increased to 6.25 mg twice daily. If heart rate < 55 beats/min, systolic blood pressure < 90 mmHg, or significant adverse reactions occur, the dose is reduced to 6.25 mg once daily; intolerable cases discontinue medication and are recorded as adverse events. Maximum dose: 12.5 mg/day (25 mg/day may be considered for patients with persistent hypertension after physician evaluation, with close blood pressure monitoring). During the first 3 months of dose adjustment, heart rate and blood pressure are checked monthly; after dose stabilization, they are checked every 3 months. Medication adherence is monitored via telephone follow-up.
  Arms: Carvedilol group

SUMMARY:
Cirrhosis is a serious liver disease where scar tissue replaces healthy liver tissue, often leading to portal hypertension-a condition where blood pressure in the liver's blood vessels rises. A life-threatening complication of this is variceal bleeding, which happens when swollen veins (varices) in the esophagus or stomach rupture. Around 30% of patients die during their first variceal bleeding episode, and 60-70% of survivors face a high risk of rebleeding, making secondary prevention crucial for improving outcomes.

Current guidelines recommend combining non-selective beta-blockers (a type of blood pressure medication) with endoscopic ligation (a procedure to tie off swollen veins) as the first-line treatment to prevent recurrent variceal bleeding. Propranolol is a commonly used non-selective beta-blocker, but it only works for 30-50% of patients by effectively reducing liver vein pressure. Carvedilol, a newer generation of this type of drug, is more potent at lowering liver vein pressure and is recommended for preventing first-time variceal bleeding. However, there is limited research on its effectiveness and safety for preventing recurrent bleeding, and concerns exist that it may cause low blood pressure, which could worsen conditions like ascites (fluid buildup in the abdomen) in some patients.

This study aims to answer a key question: Is combining endoscopic treatment with carvedilol more effective and safe than combining endoscopic treatment with propranolol for preventing recurrent bleeding in cirrhosis patients who have already experienced variceal bleeding? The research hypothesis is that carvedilol will reduce the rate of recurrent bleeding more effectively than propranolol when both are used alongside endoscopic treatment, while having a similar or acceptable safety profile.

This is a single-center randomized controlled trial conducted by the First Affiliated Hospital of Air Force Medical University, lasting 3 years (from October 2025 to October 2028). The investigators plan to recruit 350 eligible patients, aged 18-75, who have been diagnosed with cirrhosis, have a history of variceal bleeding (with the most recent episode 6-30 days before enrollment), and voluntarily agree to participate and complete follow-up. These patients will be randomly divided into two groups in a 1:1 ratio. Both groups will receive endoscopic treatment first; one group will then take propranolol, and the other will take carvedilol, with dosage adjustments based on their heart rate, blood pressure, and tolerance.

Throughout the study, the investigators will closely monitor patients for recurrent bleeding (the main measure of effectiveness) and other outcomes like disease progression, death, new or worsening ascites, liver encephalopathy (brain dysfunction due to liver disease), and changes in quality of life. The investigators will also track side effects of the drugs and complications from the endoscopic procedure to assess safety.

The results of this study will help clarify whether carvedilol can become a better choice than propranolol for preventing recurrent variceal bleeding, providing more reliable treatment guidance for cirrhosis patients and potentially improving their survival rates and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cirrhosis (based on previous liver biopsy or typical clinical features) with a history of variceal bleeding, and the most recent bleeding occurred 6-30 days before enrollment
* Aged 18-75 years (based on ID card age on the enrollment date)
* Voluntarily signs the informed consent form and can cooperate with full-course follow-up and related examinations

Exclusion Criteria:

* Non-cirrhotic portal hypertension (eg:Budd-Chiari syndrome, extrahepatic portal vein obstruction, idiopathic portal hypertension)
* Contraindications to non-selective beta-blockers (NSBBs) (eg:asthma, insulin-dependent diabetes mellitus, peripheral vascular disease)
* Malignant tumors (including hepatocellular carcinoma) or other life-shortening diseases (expected survival<1 year), including severe cardio-cerebrovascular diseases (eg:severe heart failure, bedridden status after cerebral infarction, cerebral hemorrhage), end-stage renal disease (requiring dialysis), severe pulmonary diseases (eg:acute exacerbation of chronic obstructive pulmonary disease, pulmonary fibrosis)etc
* Previous shunt or devascularization surgery, oral NSBBs, and/or endoscopic treatment for preventing recurrent variceal bleeding
* Pregnant or lactating women (female subjects must undergo a pregnancy test before enrollment; positive cases are excluded; lactating women can only enroll after stopping breastfeeding)
* Allergies to carvedilol, propranolol, or endoscopic treatment-related drugs (eg:local anesthetics, tissue adhesives)
* Severe hepatic and renal insufficiency: Child-Pugh class C with a score > 12, or MELD score > 30; serum creatinine > 221 μmol/L (2.5 mg/dl) with estimated glomerular filtration rate (eGFR) < 30 ml/(min·1.73m²)
* Severe coagulation disorders: prothrombin time (PT) prolonged by > 10 seconds, or international normalized ratio (INR) > 2.5 without effective correction measures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
All-cause recurrent bleeding | Up to 12 months
  All-cause rebleeding is the primary efficacy endpoint of this trial (per Baveno V consensus), referring to recurrent bleeding (melena or hematemesis) in cirrhotic portal hypertension patients with prior variceal bleeding-regardless of the new bleeding cause. It is defined by any of the following: hospitalization for bleeding, need for blood transfusion, hemoglobin decrease ≥ 3 g/dl, or death within 6 weeks of recurrence. Timing-wise, early rebleeding occurs 72 hours-6 weeks after initial bleeding control, and delayed rebleeding after 6 weeks. This indicator reflects the study treatments' (endoscopic ligation + carvedilol/propranolol) preventive effect on all bleeding events in cirrhotic patients.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Air Force Medical University, Xi'an, China

IPD SHARING:
Plan to Share IPD: No